CLINICAL TRIAL: NCT05874284
Title: The Effect of Prolotherapy in the Care of Pressure Injuries: A Randomized Controlled Study
Brief Title: The Effect of Prolotherapy in the Care Process of Pressure Injuries
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Rukiye Kokkiz, Research Assistant, Fenerbahce University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 22.2022fbu
Record Dates: First submitted 2023-05-13; First posted 2023-05-24 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Pressure Ulcer
Keywords: pressure injury; proliferative; wound care
MeSH Terms: conditions — Pressure Ulcer | interventions — succinylated gelatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The nasopharyngeal suction with positive pressure method was employed in the sample group. In this method, the infant's head is turned to the side, 1-2 ml of PS is injected into the nostril with a syringe, and then positive pressure is exerted with the help of the end of the oxygen hose from the same nostril, with oxygen or air supply at 5-8 lt/min (if the baby requires oxygen, using an oxygen source) and the nasopharyngeal secretions are removed from the nostril into which PS has been not injected. The oxygen hose is held one centimetre away from the infant's nostril. The researchers prepared a guideline for nasopharyngeal suction with positive pressure based on the literature.
  Interventions: Drug: Gelofusin
- conroul group (No Intervention): The nasopharyngeal suction with negative pressure method was employed in the control group in this study. In this method, the nasal secretions were softened with 1-2 ml of physiological saline (PS), and then negative pressure suction was performed using a pine-tipped suction set. In the literature, neonatal aspiration pressure is defined as 60-100 mmHg. In this study, the suction pressure was kept between 60 and 80 mmHg, and no suction lasted for more than 15 seconds.

INTERVENTIONS:
Drug: Gelofusin — In the experimental group, the wound will be washed with gelofusine as prolotherapy, and the wound will be closed with sterile sponge and fixative tape. In the control group, the wound will be covered with sterile sponge and fixative tape by washing with physiological saline.
  Other Names: there is no other name
  Arms: Experimental group

SUMMARY:
The goal of this [type of study: randomized controlled clinical trial] is to [Determining the effect of prolotherapy use on the wound care process]. The main question it aims to answer is:

• [The use of proliferative substances in the care of 1st, 2nd and 3rd stage pressure injuries has a positive effect on the wound healing period].

Participants will [in patients with pressure injuries, wound irrigation with saline and wound irrigation with gelofusin were applied]. Researchers will compare [depth, length and width of the wound].

DETAILED DESCRIPTION:
In the study, wound irrigation with saline and wound irrigation with gelofusin will be applied to patients with pressure injuries.

Cleaning of the wound can be done with gases moistened with saline, or irrigation method can be applied with the help of an injector. Sufficient pressure can be provided with an 18G needle attached injector. Irrigation with 50-100cc saline per square centimeter is recommended.

In the experimental group, the wound will be washed with gelofusine as prolotherapy, and the wound will be closed with sterile sponge and fixative tape. In the control group, the wound will be covered with sterile sponge and fixative tape by washing with physiological saline. This process will be repeated 2 times a day and will be repeated and observed for 3 days in line with the literature.

In this study, while the wound is irrigated, the solution will first be drawn into a 50 cc syringe and prepared. A protective cover will be used to prevent the sterile sponge, fixation tape, gloves and solution required for dressing from contaminating the patient bed. The patient will be given an appropriate position according to the location of the wound. The needle of the syringe containing the solution will be removed and kept at a distance of 3 cm from the wound area, and the solution will be slowly poured over the entire wound. When the irrigation process is finished, the wound area will be dried and the wound will be closed with sterile sponge.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 1st, 2nd and 3rd stage pressure injuries
* Patients over 18 years of age
* Patients who volunteered to participate in the study

Exclusion Criteria:

* Patients without 1st, 2nd and 3rd stage pressure injuries
* Patients under 18 years of age
* Patients who did not volunteer to participate in the study
* Patients allergic to gelofusin solution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
wound healing time | 3 days
  The change in wound healing time will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Fenerbahce University, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No